CLINICAL TRIAL: NCT03397576
Title: A Randomized Controlled Trial of a Medication Adherence Intervention (ATHENA-I) to Increase Adherence to Antiretroviral Therapy Among HIV-Infected Prisoners in Indonesia
Brief Title: Adherence Through Home Education and Nursing Assessment, Indonesia
Acronym: ATHENA-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Indonesia University (Other)
Responsible Party: Principal Investigator, Gabriel John Culbert, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-0196
Record Dates: First submitted 2017-09-26; First posted 2018-01-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: HIV/AIDS; Medication Adherence; Substance Use
Keywords: Prisoner
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blinded to treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATHENA (Experimental): Subjects in the experimental arm will participate in monthly group medication adherence counseling sessions within prison led by a nurse and peer educator. After prison release, subjects in the experimental group will participate in four home visits during which intervention staff (nurses and peer educators working in teams) will deliver individualized medication adherence counseling based on the Freirian educational model.
  Interventions: Behavioral: ATHENA
- Control (No Intervention): Subjects in the control group will receive standard care, which includes a referral for HIV care and ART if prescribed ART within prison.

INTERVENTIONS:
Behavioral: ATHENA — Adherence Through Home Education and Nursing Assessment (ATHENA), is an evidence-based ART adherence intervention delivered in the patient's home by nurses and peer educators working in teams.
  Arms: ATHENA

SUMMARY:
Adherence to antiretroviral therapy (ART) drops sharply after prison release. Effective medication adherence training immediately before and after prison release may improve health outcomes and limit transmission of Human Immunodeficiency Virus (HIV). ATHENA (Adherence Through Home Education and Nursing Assessment) is an evidence-based medication adherence intervention, which is delivered in the patient's home by nurses and peer educators working in teams. In this study, researchers will examine the acceptability and feasibility of the ATHENA intervention through a 2-arm randomized controlled trial conducted with HIV-infected prisoners in Indonesia. Eligible subjects will be >18 years of age, HIV-infected, and may be treatment-experienced or treatment-naive. Subjects randomized to the intervention arm will participate in monthly medication adherence counseling sessions within prison and home visits up to four months after prison release. Subjects randomized to the control arm will receive standard care, which includes a referral for HIV care after prison release. The primary endpoint is the proportion of subjects demonstrating ART adherence >90% at 3 months after prison release. Secondary endpoints are: 1) retention in HIV care, 2) ART initiation, 3) HIV- RNA viral load, 4) CD4+ T-cell count, 5) quality of life, 6) hospitalization, 6) substance use and sexual risk behaviors at 3 months after prison release.

DETAILED DESCRIPTION:
The acceptability and feasibility of the adapted ATHENA intervention will be assessed through a 2-arm randomized controlled trial conducted in two phases with HIV-infected prisoners recruited from 2 correctional facilities in Jakarta, Indonesia.

Phase 1: HIV+ prisoners who are already aware of their status will be recruited through prison clinics and randomized to receive either the adapted ATHENA intervention or standard care as a control. Uniform data collection at baseline will include measures of ART adherence, HIV stigma, and drug dependence and CD4+ T-cell and viral load testing.

Phase 2: Subjects receiving the ATHENA intervention will participate in monthly medication adherence counseling sessions within prison, and home visits up to four months after prison release, during which intervention staff (nurses and peer educators working in teams) will deliver individualized medication adherence counseling based on the Freirian educational model.

Phase 3: Participants in both groups will be followed for 12 months after prison release, and asked to complete monthly study visits to evaluate primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection documented by a rapid HIV test or any licensed ELISA test; and confirmed by another test using a different method, including but not limited to rapid HIV tests, Western Blot, HIV culture, HIV antigen, or HIV pro-viral DNA at any time prior to study entry; and aware of HIV status
* age ≥ 18 years
* Karnofsky performance score >40
* conversant in Bahasa Indonesia

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Adherence to antiretroviral therapy (ART) | 3 months after prison release
  Adherence to antiretroviral therapy >90%

SECONDARY OUTCOMES:
Retention in HIV care | 3 months after prison release
  Being seen by an HIV care provider
ART initiation | 3 months after prison release
  Having initiated or continued ART
Viral load | 3 months after prison release
  HIV-RNA viral load
CD4+ T-cell count | 3 months after prison release
  CD4+ T-cell count
Quality of life | 3 months after prison release
  Quality of life as assessed by WHO Quality of Life scale
Hospitalization | 3 months after prison release
  Frequency of hospitalization or emergency department visits
Drug and Sexual Risk Behaviors | 3 months after prison release
  Frequency of drug and sexual risk behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel J Culbert, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Indonesia, Depok, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided